CLINICAL TRIAL: NCT03580122
Title: Does Arginine Enhance Galactose Oxidative Capacity in Classic Galactosemia: A Pilot Study
Brief Title: The Effect of Arginine on Classic Galactosemia
Acronym: ARGALT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Ana Coelho, Coordinating Investigator, Academisch Ziekenhuis Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL49929.068.17
Record Dates: First submitted 2018-06-05; First posted 2018-07-09 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Classic Galactosemia
MeSH Terms: conditions — Galactosemias | interventions — arginine aspartate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asparten (Experimental): Asparten (arginine aspartate) 5000mg/10mL 3x/day
  Interventions: Drug: Arginine Aspartate

INTERVENTIONS:
Drug: Arginine Aspartate — Asparten

SUMMARY:
Rationale: Classic galactosemia is a rare inherited metabolic disease that presents in neonatal patients with a life-threatening multi-organ toxic syndrome. Although the current standard of care - a galactose-restricted diet - quickly relieves the severe neonatal clinical picture, it fails to prevent brain and gonadal sequelae. There is a need for new therapeutic strategies.

As arginine is an amino acid that is therapeutically widely used with no side effects described, we propose to use it in a pilot-clinical study. We aim to evaluate the effects of arginine in classic galactosemia patients, in order to determine its potential therapeutic role in this disease.

Objective: To evaluate the possible effect of arginine on the whole body galactose oxidative capacity in classic galactosemia patients.

Study design: Interventional pilot-clinical study with pre-post single arm design.

Study population: We aim to include 5 classic galactosemia adult patients homozygous for the p.Q188R mutation.

Intervention: All participants will receive arginine in the form of Asparten ® (arginine aspartate) during 1 month, by oral administration.

The main study parameter is whole body galactose galactose oxidative capacity.

ELIGIBILITY:
Inclusion Criteria:

* Classic galactosemia patient homozygous for the p.Q188R mutation, diagnosed by GALT enzyme activity assay and GALT gene mutation analysis
* Eighteen years of age or older
* Capable of giving informed consent

Exclusion Criteria:

* Urea cycle disorders (assessed by post prandial amino acid profile in blood)
* Increased level of plasma uric acid
* Patients experiencing acute illness of classic galactosemia
* Pregnant women (or considering getting pregnant) or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
whole body galactose oxidative capacity | 6 hours
  Whole body galactose oxidative capacity is breathing test that quantifies [1-13C]-galactose conversion into 13CO2, thus allowing to delineate the exact extent of impaired galactose metabolism, providing clear information on a patient's ability to oxidize galactose.

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Ziekenhuis Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Haskovic M, Derks B, van der Ploeg L, Trommelen J, Nyakayiru J, van Loon LJC, Mackinnon S, Yue WW, Peake RWA, Zha L, Demirbas D, Qi W, Huang X, Berry GT, Achten J, Bierau J, Rubio-Gozalbo ME, Coelho AI. Arginine does not rescue p.Q188R mutation deleterious effect in classic galactosemia. Orphanet J Rare Dis. 2018 Nov 26;13(1):212. doi: 10.1186/s13023-018-0954-8. PMID 30477550